CLINICAL TRIAL: NCT02199548
Title: The Good Patient Study
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GPS14
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Solid Tumor; Hematological Malignancies; Brain Tumor
Keywords: Adolescent; Decision-making; Social network
MeSH Terms: conditions — Hematologic Neoplasms; Brain Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Participants: All enrolled participants will take part in a face-to-face interview.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — This study involves teen participants taking part in one private interview with the study team. Interviews last less than one hour and are scheduled at the participant's convenience. Interviews will be audio/digital recorded. Participants may answer any or all of the questions.

SUMMARY:
Adolescents with cancer weigh multiple influences in medical decision-making, including their own best interest, the perceived wishes of family members, and the interpreted preferences of the health care team. Parents of children with cancer often describe themselves as trying to be a good parent in making decisions in the child's best interest. Adolescents with cancer often describe themselves as trying to be a good patient and good child in making decisions in accord with how they believe a good patient and good child would decide.

Among the challenges of caring for adolescents is the reality that the formative relational influences in adolescents' decision-making are both complex and unique due to adolescent patients' social networks and relational roles. Delineating adolescents' definitions of being a good patient, a good child, a good sibling, and a good friend may enable the care team to better understand the formative decisional influences relevant to adolescents with cancer. Expanding knowledge about the decision making constructs relevant to adolescents with cancer and recognizing the role of these social constructs in medical interactions has the potential for development of a comprehensive care model that methodically evaluates the self-assessed decision making influences and needs of adolescents at various stages in oncology care.

This qualitative construct-defining study represents an initial step in the development of enhanced interventions for improved psychosocial support in this vulnerable population.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* Describe the ways relationships and social interactions may factor into adolescent study participants' approach to decisions;
* By reports from adolescents with cancer, identify behaviors from members of the study participants' social network that would be helpful to adolescents in fulfilling their preferred role in medical decision-making and achieving the desired level of participation in medical decision-making;
* Identify adolescent participants' preferred role in medical decision making.

SECONDARY OBJECTIVES:

* Develop definitions of being a "good" patient, child, sibling, and friend from adolescent participant reports (will also welcome the study participant to self-declare any additional relational constructs they may wish to report);
* Describe how the adolescent study participant believes his or her "good" patient, child, sibling, and friend definition may have changed over time;
* Describe the self-assessed positive and negative aspects of trying to achieve the meanings of the "good" patient, child, sibling, and friend constructs from adolescent participant reports;
* Describe the actions of members of the study participant's social network which may help the study participant reach his/her definition of being a "good" patient, child, sibling, and friend.

Participants will participate in a one-time voice-recorded, face-to-face interview consisting of open-ended questions. Completion of the interview is expected to take less than one hour.

The qualitative interview consists of thirty open-ended questions for participants with no siblings and thirty-eight open-ended questions for participants who have siblings. Questions will be audio-recorded, face-to-face semi-structured in-depth interview format. Health information will also be collected from medical records.

Expected accrual is 100 participants, 50 at each participating site. Accrual will be halted when the study reaches qualitative theme saturation. For this study, saturation will occur when three consecutive interviews fail to raise a new theme.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 12 and 19 years of age at the time of enrollment.
* Participants must have primary care team approval to participate.
* Participants must be English-speaking.
* Participants must carry an oncologic diagnosis.
* Participants must be within four months of initial oncologic diagnosis or within four months of relapse/recurrent disease.

Exclusion Criteria:

* This study lacks any exclusion related to pregnancy (an Institutional Review Board requirement for enrollment of females who are capable of becoming pregnant), lactation or plans to become pregnant and lacks any exclusion of males fathering children while on study.
* Patients who, in the opinion of their physician, are not capable mentally or verbally of participating in the interview, will be excluded from the study.

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be teens who are patients at St. Jude Children's Research Hospital and meet the criteria for study enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Factors contributing to decision-making | Once, at enrollment
  Describe the ways relationships and social interactions may factor into adolescent study participants' approach to decisions.
Behaviors that make a positive impact on decision-making | Once, at enrollment
  By reports from adolescents with cancer, identify behaviors from members of the study participants' social network that would be helpful to adolescents in fulfilling their preferred role in medical decision-making and achieving the desired level of participation in medical decision-making.
Preferred decision-making role | Once, at enrollment
  Identify adolescent participants' preferred role in medical decision making.

CONTACTS AND LOCATIONS:
Overall Officials: Meaghann Weaver, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - Children's National Health System, Washington D.C., District of Columbia
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols